CLINICAL TRIAL: NCT04904614
Title: Evaluation of the Tolerability and Clinical Effectiveness of Letermovir in Heart Transplantation
Brief Title: Letermovir Use in Heart Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00001538
Record Dates: First submitted 2021-05-10; First posted 2021-05-27 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Cytomegalovirus Disease; Cytomegalovirus Infections; Heart Transplant Infection; Antiviral Toxicity; Neutropenia
Keywords: cytomegalovirus, letermovir, heart transplantation
MeSH Terms: conditions — Cytomegalovirus Infections; Neutropenia | interventions — letermovir

STUDY DESIGN:
Intervention Model Description: Open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- single arm (Other): Letermovir 480 mg daily for cmv prophylaxis
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Open label trial of the licensed drug, letermovir, in a population of heart transplant recipients for which it is not yet licensed
  Other Names: Prevymis

SUMMARY:
This is an open label trial in which letermovir will be given as prophylaxis for the prevention of cytomegalovirus (CMV) infection and disease to all heart transplants who are at risk for cytomegalovirus. The study will compare a 30 patient prospective cohort to a retrospective cohort of 374 heart transplant recipients for the rates of neutropenia. In addition, the tolerability of letermovir will be assessed in this population.

DETAILED DESCRIPTION:
This open label trial will follow 30 heart transplant recipients at Tufts Medical Center who will receive letermovir in a dose of 480 mg daily for either 3 or 6 months depending on the CMV risk category, and who will be followed for one year. Comparison will be made to a cohort of heart transplant recipients as historical controls in a recently presented study (Chow, J, et al ISHLT 2021). Standard follow up will be provided as if the patients were receiving valganciclovir prophylaxis. Post prophylaxis T cell immunity to all subjects enrolled will be tested. Clinical outcomes are detailed below.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18-70 will be eligible for participation
2. Written informed consent and able to participate with follow up
3. Heart transplant recipients who are not Cytomegalovirus (CMV) donor negative and CMV recipient negative (CMV D-/R-)
4. Not enrolled in competing clinical trials

Exclusion Criteria:

1. Dual heart and kidney transplant recipients
2. Patients who do not survive 72 hours post transplant
3. HIV infection
4. Patients with creatinine clearance less than 10 ml per min at time of enrollment
5. Hypersensitivity to letermovir
6. On continuous veno-venous hemofiltration or renal dialysis at the time of enrollment
7. Received a previous solid organ transplant or stem cell transplant.
8. Has Child Pugh Class C severe hepatic insufficiency at screening.
9. Has both moderate hepatic insufficiency AND moderate to severe renal insufficiency at screening.

   Note: Moderate hepatic insufficiency is defined as Child Pugh Class B; moderate to severe renal insufficiency is defined as Creatine Clearance <50 mL/min, as calculated by the Cockcroft-Gault equation (as above), respectively.
10. Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy.
11. Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through at least 90 days following cessation of study therapy.
12. Is expecting to donate eggs or sperm starting from the time of consent through at least 90 days following cessation of study therapy.
13. Has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or put the participant at undue risk, as judged by the investigator, such that it is not in the best interest of the participant to participate in this study.
14. Has exclusionary laboratory value at screening, as listed in Table 1. Table 1 Laboratory Exclusion Criteria Laboratory Assessment Exclusionary Value

    Hemoglobin <8 g/dL Platelets <25,000 cells/µL Absolute neutrophil count <1,000 cells/µL Total bilirubin >2.5 × ULN ALT >5 × ULN AST >5 × ULN

    ALT = alanine aminotransferase; AST = aspartate aminotransferase; CMV = cytomegalovirus; IgG = immunoglobulin G; ULN = upper limit of normal
15. Is currently participating or has participated in a study with an unapproved investigational compound or device within 28 days, or 5× half-life of the investigational compound (excluding monoclonal antibodies), whichever is longer, of initial dosing on this study. Participants previously treated with an investigational monoclonal antibody will be eligible to participate after a 150-day washout period.

    Note: Investigational regimens involving combinations of approved agents are not permitted. Other non-interventional or other observational studies are allowed.
16. Has previously participated in this study or any other study involving letermovir.
17. Has previously participated or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent, or is planning to participate in a study of a CMV vaccine or another CMV investigational agent during the course of this study.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotton CN, Kumar D, Caliendo AM, Huprikar S, Chou S, Danziger-Isakov L, Humar A; The Transplantation Society International CMV Consensus Group. The Third International Consensus Guidelines on the Management of Cytomegalovirus in Solid-organ Transplantation. Transplantation. 2018 Jun;102(6):900-931. doi: 10.1097/TP.0000000000002191. PMID 29596116
- [Background] Snydman DR. Epidemiology of infections after solid-organ transplantation. Clin Infect Dis. 2001 Jul 1;33 Suppl 1:S5-8. doi: 10.1086/320897. PMID 11389515
- [Background] Marty FM, Ljungman P, Chemaly RF, Maertens J, Dadwal SS, Duarte RF, Haider S, Ullmann AJ, Katayama Y, Brown J, Mullane KM, Boeckh M, Blumberg EA, Einsele H, Snydman DR, Kanda Y, DiNubile MJ, Teal VL, Wan H, Murata Y, Kartsonis NA, Leavitt RY, Badshah C. Letermovir Prophylaxis for Cytomegalovirus in Hematopoietic-Cell Transplantation. N Engl J Med. 2017 Dec 21;377(25):2433-2444. doi: 10.1056/NEJMoa1706640. Epub 2017 Dec 6. PMID 29211658
- [Background] Goldner T, Hewlett G, Ettischer N, Ruebsamen-Schaeff H, Zimmermann H, Lischka P. The novel anticytomegalovirus compound AIC246 (Letermovir) inhibits human cytomegalovirus replication through a specific antiviral mechanism that involves the viral terminase. J Virol. 2011 Oct;85(20):10884-93. doi: 10.1128/JVI.05265-11. Epub 2011 Jul 13. PMID 21752907
- [Background] Kaul DR, Stoelben S, Cober E, Ojo T, Sandusky E, Lischka P, Zimmermann H, Rubsamen-Schaeff H. First report of successful treatment of multidrug-resistant cytomegalovirus disease with the novel anti-CMV compound AIC246. Am J Transplant. 2011 May;11(5):1079-84. doi: 10.1111/j.1600-6143.2011.03530.x. PMID 21521474
- [Background] Marschall M, Stamminger T, Urban A, Wildum S, Ruebsamen-Schaeff H, Zimmermann H, Lischka P. In vitro evaluation of the activities of the novel anticytomegalovirus compound AIC246 (letermovir) against herpesviruses and other human pathogenic viruses. Antimicrob Agents Chemother. 2012 Feb;56(2):1135-7. doi: 10.1128/AAC.05908-11. Epub 2011 Nov 21. PMID 22106211
- [Background] Lischka P, Hewlett G, Wunberg T, Baumeister J, Paulsen D, Goldner T, Ruebsamen-Schaeff H, Zimmermann H. In vitro and in vivo activities of the novel anticytomegalovirus compound AIC246. Antimicrob Agents Chemother. 2010 Mar;54(3):1290-7. doi: 10.1128/AAC.01596-09. Epub 2010 Jan 4. PMID 20047911
- [Background] Giulieri S, Manuel O. QuantiFERON(R)-CMV assay for the assessment of cytomegalovirus cell-mediated immunity. Expert Rev Mol Diagn. 2011 Jan;11(1):17-25. doi: 10.1586/erm.10.109. PMID 21171917
- [Background] Ljungman P, Boeckh M, Hirsch HH, Josephson F, Lundgren J, Nichols G, Pikis A, Razonable RR, Miller V, Griffiths PD; Disease Definitions Working Group of the Cytomegalovirus Drug Development Forum. Definitions of Cytomegalovirus Infection and Disease in Transplant Patients for Use in Clinical Trials. Clin Infect Dis. 2017 Jan 1;64(1):87-91. doi: 10.1093/cid/ciw668. Epub 2016 Sep 28. PMID 27682069
- [Background] Gardiner BJ, Nierenberg NE, Chow JK, Ruthazer R, Kent DM, Snydman DR. Absolute Lymphocyte Count: A Predictor of Recurrent Cytomegalovirus Disease in Solid Organ Transplant Recipients. Clin Infect Dis. 2018 Oct 15;67(9):1395-1402. doi: 10.1093/cid/ciy295. PMID 29635432
- [Background] Arbo MD, Snydman DR. Influence of blood culture results on antibiotic choice in the treatment of bacteremia. Arch Intern Med. 1994 Dec 12-26;154(23):2641-5. doi: 10.1001/archinte.1994.00420230024004. PMID 7993147
- [Background] George MJ, Snydman DR, Werner BG, Griffith J, Falagas ME, Dougherty NN, Rubin RH. The independent role of cytomegalovirus as a risk factor for invasive fungal disease in orthotopic liver transplant recipients. Boston Center for Liver Transplantation CMVIG-Study Group. Cytogam, MedImmune, Inc. Gaithersburg, Maryland. Am J Med. 1997 Aug;103(2):106-13. doi: 10.1016/s0002-9343(97)80021-6. PMID 9274893

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in the historical control arm were not considered enrolled in this study.
Groups:
- Single Arm: Letermovir 480 mg daily for cytomegalovirus (CMV) prophylaxis
- Historical Controls: Retrospectively collected historical controls who received valganciclovir for CMV prophylaxis; not enrolled in current study
  A total of 204 CMV D+/R- and CMV R+ patients on valganciclovir for CMV prophylaxis formed our historical control group of adult heart transplant (HT) recipients at Tufts Medical Center from January 2004 to December 2017 who were followed for one-year post-HT for development of neutropenia, as well as infection, rejection, and survival.
  Chow JKL, Ruthazer R, Boucher HW, Vest AR, DeNofrio DM, Snydman DR: Factors associated with neutropenia post heart transplantation. Transpl Infect Dis 2021;23:e13634.
Period: Overall Study
Arm/Group | Single Arm | Historical Controls
Started | 32 | 204
Completed | 32 | 204
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: historical controls not enrolled in current study
Groups:
- Intervention Arm: Letermovir 480 mg daily for cmv prophylaxis
  Letermovir: Open label trial of the licensed drug, letermovir, in a population of heart transplant recipients for which it is not yet licensed
- Historical Controls: A total of 204 CMV D+/R- and CMV R+ patients on valganciclovir for CMV prophylaxis formed our historical control group of adult HT recipients at Tufts Medical Center from January 2004 to December 2017 who were followed for one-year post-HT for development of neutropenia, as well as infection, rejection, and survival.
  These patients were NOT enrolled in current study.
  Chow JKL, Ruthazer R, Boucher HW, Vest AR, DeNofrio DM, Snydman DR: Factors associated with neutropenia post heart transplantation. Transpl Infect Dis 2021;23:e13634.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Historical Controls | Total
Number analyzed (Participants) | 32 | 204 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12) | 53 (12) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 60 | 66
  Male | 26 | 144 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 24 | 29
  Not Hispanic or Latino | 27 | 180 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 15 | 19
  White | 27 | 184 | 211
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 204 | 236
CMV Donor IgG seropositive/Recipient IgG seronegative (CMV D+/R-) [Count of Participants; unit: Participants] — CMV Donor IgG positive serostatus/CMV Recipient IgG negative serostatus = CMV D+R-
  Participants | 19 | 85 | 104

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Neutropenia Compared to Historical Controls
Description: We will count the number of patients with neutropenia seen over one year and calculate the proportion who become neutropenic. A comparison group of historic controls from a similar population is available for comparison. We know the control group has a 30% likelihood of becoming neutropenic at one year.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm | Historical Controls
Number analyzed (Participants) | 32 | 204
Participants | 0 | 30
Statistical Analysis 1: Comparison: Single Arm vs Historical Controls; Test type: Superiority; p = 0.02, Fisher Exact

2. Secondary Outcome: Rate of CMV Infection in Letermovir Recipients Compared to Historical Controls
Description: Number of patients who develop CMV infection, comparison will be made to historic control group who were taking valganciclovir for CMV prophylaxis
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Historical Control Group: A total of 204 CMV D+/R- and CMV R+ patients on valganciclovir for CMV prophylaxis formed our historical control group of adult HT recipients at Tufts Medical Center from January 2004 to December 2017 who were followed for one-year post-HT for development of neutropenia, as well as infection, rejection, and survival.
  These patients were NOT enrolled in current study.
  Chow JKL, Ruthazer R, Boucher HW, Vest AR, DeNofrio DM, Snydman DR: Factors associated with neutropenia post heart transplantation. Transpl Infect Dis 2021;23:e13634.
Arm/Group | Single Arm | Historical Control Group
Number analyzed (Participants) | 32 | 204
Participants | 11 | 50
Statistical Analysis 1: Comparison: Single Arm vs Historical Control Group; Test type: Superiority; p = 0.13, Chi-squared

3. Secondary Outcome: Rate of Opportunistic Infections in Letermovir Arm Compared to Historical Controls
Description: Number of patients who develop an opportunistic infection
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm | Historical Controls
Number analyzed (Participants) | 32 | 204
Participants | 3 | 25
Statistical Analysis 1: Comparison: Single Arm vs Historical Controls; Test type: Superiority; p = 0.6, Fisher Exact

4. Secondary Outcome: Tolerability and Compliance of Letermovir
Description: Number of patients with adverse events will be collected using a data questionnaire, and examination of lab data, need for subsequent hospitalization.
  There is no comparator group for this purely descriptive outcome.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 32
Participants | 0

5. Secondary Outcome: Use of Granulocyte Colony Stimulation Factor (GCSF) in Letermovir Recipients Compared to Historical Controls
Description: Comparison of Proportions
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm | Historical Controls
Number analyzed (Participants) | 32 | 204
Participants | 9 | 58
Statistical Analysis 1: Comparison: Single Arm vs Historical Controls; Test type: Superiority; p = 0.97, Chi-squared

6. Secondary Outcome: Measure of CMV Specific T Cell Immunity in Letermovir Recipients
Description: Single measurement of specific T-cell immune function to CMV. There is no comparator arm for this outcome because this test did not exist at time of historical controls.
  This is a measure of CMV specific T-cell immunity based on a commercial assay that yields one of 3 results: positive (CMV T-cell function is measured), indeterminate, negative (CMV T-cell function is not measured). A positive T-cell test is considered a better outcome.
Time Frame: single time point measured within 2 weeks after completion of prophylaxis therapy, at either 3 months or 6 months, depending on duration of prophylaxis
Population: 3 missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 29
Participants
  positive CMV T-cell test | 20
  negative CMV T-cell test | 4
  Indeterminate CMV T-cell test | 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Single Arm | Historical Controls
All-Cause Mortality (participants affected / at risk) | 0/32 | 10/204
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/204
Other Adverse Events (participants affected / at risk) | 0/32 | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT04904614/Prot_SAP_000.pdf